CLINICAL TRIAL: NCT03005288
Title: A Randomized, Subject- and Investigator-blinded, Placebo Controlled Study to Assess the Safety, Pharmacokinetics and Efficacy of Intravenous Bimagrumab in Overweight and Obese Patients With Type 2 Diabetes
Brief Title: Safety, Pharmacokinetics and Efficacy of Bimagrumab in Overweight and Obese Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBYM338X2211
Record Dates: First submitted 2016-12-24; First posted 2016-12-29 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; obesity; DXA; MRI
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — bimagrumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BYM338 10 mg/kg (Experimental): Bimagrumab (BYM338) 10 mg/kg up to maximum 1200 mg, every 4 weeks until week 44 (12 doses)
  Interventions: Drug: BYM338 10 mg/kg
- Placebo (Placebo Comparator): Placebo, every 4 weeks until week 44 (12 doses)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BYM338 10 mg/kg — intravenous infusion every four weeks
  Other Names: Bimagrumab
  Arms: BYM338 10 mg/kg
Other: Placebo — intravenous infusion every four weeks
  Arms: Placebo

SUMMARY:
This study assessed the safety, pharmacokinetics and efficacy of bimagrumab when administered in overweight and obese patients with type 2 diabetes

DETAILED DESCRIPTION:
A non-confirmatory, randomized, subject and investigator blinded, placebo controlled, parallel-arm study, investigating a 48-week treatment period with i.v. bimagrumab 10 mg/kg in overweight and obese subjects with type 2 diabetes.

Participants were randomized and assigned to one of the following 2 treatment arms in a ratio of 1:1:

Arm 1: Bimagrumab 10 mg/kg up to maximum 1200 mg, every 4 weeks (12 doses) until week 44.

Arm 2: Placebo, every 4 weeks (12 doses) until week 44.

The study consisted of a screening baseline period of 3 weeks, treatment period of 48 weeks and then a follow-up period of 8 weeks.

Treatment period visits were scheduled every 4 weeks until week 44. Administration of bimagrumab or placebo was done via an i.v. infusion over 30 minutes followed by flushing for 15 minutes. Subjects were asked to return to the Investigator site for dosing approximately every 4 weeks during the treatment period. During those visits, subjects were evaluated for safety, tolerability, PK and efficacy. The treatment period ended approximately 4 weeks after the last dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with HbA1c between 6.5% and 10% at screening with stable treatment for 3 months prior to randomization
* On one of the following anti-diabetes regimens with stable treatment for approximately 3 months prior to randomization: 1) metformin monotherapy; 2) DPP4 inhibitor agent monotherapy; 3) combination therapy of metformin and DPP4 inhibitor agent; 4) no anti-diabetes therapy.
* Body Mass Index of 28 to 40 kg/m2 at screening
* Body weight between 65 and 140 kg at screening

Exclusion Criteria:

* Women of child-bearing potential unless they are using highly effective methods of contraception
* Diabetes other than Type 2 such as Type 1 diabetes, surgically induced diabetes, "brittle" type 2 diabetes as per investigator judgement, history of severe hypoglycemic episodes in the year preceding screening or hypoglycemic unawareness
* History of clinically significant arrythmias, heart failure, unstable angina, myocardial infarction or stroke, coronary artery bypass graft surgery, or percutaneous coronary intervention, deep vein thrombosis/pulmonary embolism, valve disorders or defects, pulmonary hypertension within 6 months of screening or 1 year for drug-eluting stents
* Tachycardia
* Use of anti-obesity medications, nutritional supplements or over the counter products for weight loss within 3 months of screening
* Use of medications known to induce weight gain such as some anti-convulsant and psychotropic medications within 3 months of screening
* Any chronic active infection (e.g., HIV, Hepatitis B or C, tuberculosis, etc) or has received anti-HCV treatments within the previous 6 months.
* Uncontrolled thyroid disease. Stable euthyroid patients on stable thyroid replacement therapy for at least 3 months of screening are allowed.
* Abnormal liver function tests such as SGOT, SGPT, alkaline phosphatase, or serum bilirubin, or abnormal lipase and/or amylase.
* Known history or presence of severe active acute or chronic liver disease (e.g., cirrhosis).
* Uncontrolled depression
* Use of skeletal muscle anabolic agents in any form for 3 months prior to screening
* Chronic kidney disease [estimated glomerular filtration rate (GFR) < 30 mL/min];

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (7):
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Miami Lakes, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Berlin, New Jersey
  - Novartis Investigative Site, Eatontown, New Jersey
- Novartis Investigative Site, Merthyr Tydfil, Mid Glamorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Heymsfield SB, Coleman LA, Miller R, Rooks DS, Laurent D, Petricoul O, Praestgaard J, Swan T, Wade T, Perry RG, Goodpaster BH, Roubenoff R. Effect of Bimagrumab vs Placebo on Body Fat Mass Among Adults With Type 2 Diabetes and Obesity: A Phase 2 Randomized Clinical Trial. JAMA Netw Open. 2021 Jan 4;4(1):e2033457. doi: 10.1001/jamanetworkopen.2020.33457. PMID 33439265
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was completed as planned.
Pre-assignment Details: Participants were randomized to the study at 1:1 ratio to receive BYM338 10 mg/kg or placebo.
Period: Overall Study
Arm/Group | BYM338 10 mg/kg | Placebo
Started (All the participants who were assigned a randomization number.) | 39 | 39
Safety Analysis Set (All subjects that received any study drug.) | 37 | 38
Pharmacokinetics (PK) Analysis Set (All subjects who received any study drug and experienced no protocol deviations.) | 36 (One subject was excluded due to a protocol deviation.) | 0 (PK samples were only obtained and evaluated for subjects treated with BYM338.)
Pharmacodynamics (PD) Analysis Set (All subjects who received any study drug and experienced no protocol deviations.) | 36 (One subject was excluded due to a protocol deviation.) | 36 (Two subjects were excluded due to protocol deviations.)
Completed | 27 | 31
Not Completed | 12 | 8
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 5 | 0
Not completed — Protocol deviation | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 78 participants were randomized and were assigned to the respective treatment groups. Of the 78 participants, 3 withdrew from the study prior to dosing due to subject/physician decision. The remaining 75 participants underwent baseline assessments and treatment analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | BYM338 10 mg/kg | Placebo | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (7.50) | 60.2 (8.02) | 60.4 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 12 | 35
  Male | 14 | 26 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black Or African American | 6 | 9 | 15
  Race: Other | 1 | 0 | 1
  Race: White | 30 | 27 | 57
  Race: Asian | 0 | 1 | 1
  Race: Unknown | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic Or Latino | 27 | 25 | 52
  Ethnicity: Not Hispanic Or Latino | 9 | 12 | 21
  Ethnicity: Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Body Fat Mass by Dual Energy X-ray Absorptiometry (DXA) at Week 48
Description: Dual energy X-ray absorptiometry (DXA) was used to assess changes in body composition, including total fat and lean body mass (FM and LBM) and appendicular skeletal fat and muscle mass (aFM and aLBM). DXA instruments had a source that generated x-rays split into two energies which measured bone mineral mass and soft tissue from which fat and fat-free mass (or lean body mass) were estimated.
Time Frame: Baseline, Week 48
Population: Pharmacodynamic (PD) analysis set
Measure: Least Squares Mean (80% Confidence Interval); unit: kg
Arm/Group | BYM338 10 mg/kg | Placebo
Number analyzed (Participants) | 36 | 36
kg | -7.49 [-8.33 to -6.64] | -0.18 [-0.99 to 0.63]
Statistical Analysis 1: Comparison: BYM338 10 mg/kg vs Placebo; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = -7.31, 80% CI 2-sided [-8.48 to -6.14]

2. Secondary Outcome: Change From Baseline in Total Body Fat Mass by Dual Energy X-ray Absorptiometry (DXA) at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: Pharmacodynamic analysis set
Measure: Least Squares Mean (80% Confidence Interval); unit: kg
Arm/Group | BYM338 10 mg/kg | Placebo
Number analyzed (Participants) | 36 | 36
kg | -5.37 [-5.96 to -4.78] | -0.18 [-0.75 to 0.39]
Statistical Analysis 1: Comparison: BYM338 10 mg/kg vs Placebo; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = -5.19, 80% CI 2-sided [-6.01 to -4.37]

3. Secondary Outcome: Change From Baseline in HbA1c at Week 24 and 48
Description: HbA1c reflects average glucose concentrations over the past 3 months and therefore provides a useful index of the glycemic control of bimagrumab over that time period. It is a standard endpoint used to assess the glycemic efficacy of any anti-diabetic medication. HbA1c is a key glycemic parameter which correlates with reduction of risk of diabetic complications.
Time Frame: Baseline, Week 24, Week 48
Population: Pharmacodynamic analysis set
Measure: Least Squares Mean (80% Confidence Interval); unit: percentage change
Arm/Group | BYM338 10 mg/kg | Placebo
Number analyzed (Participants) | 36 | 36
percentage change
  week 24: number analyzed (Participants) | 29 | 31
  week 24 | -0.85 [-1.06 to -0.64] | 0.28 [0.08 to 0.48]
  week 48: number analyzed (Participants) | 26 | 30
  week 48 | -0.76 [-1.05 to -0.48] | 0.04 [-0.23 to 0.31]
Statistical Analysis 1: Comparison: BYM338 10 mg/kg vs Placebo; week 24; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.13, 80% CI 2-sided [-1.42 to -0.83]
Statistical Analysis 2: Comparison: BYM338 10 mg/kg vs Placebo; week 48; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Net) = -0.80, 80% CI 2-sided [-1.20 to -0.41]

4. Secondary Outcome: The Trough Observed Analyte Concentration (Ctrough) of Repeat Doses of BYM338 10 mg/kg on Day 84, 168, 252, 308 and 336
Description: The trough observed analyte concentration (Ctrough) is the concentration that is just prior to the beginning of, or at the end of, a dosing interval (μg/mL).
Time Frame: Day 84, 252, 336 at pre-dose only. Day 168, 308 at pre-dose and 45 mins post-dose
Population: Pharmacokinetics (PK) analysis set - PK samples were only obtained and evaluated for subjects treated with BYM338
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | BYM338 10 mg/kg | Placebo
Number analyzed (Participants) | 36 | 0
μg/mL
  Day 84: number analyzed (Participants) | 29 | 0
  Day 84 | 25.3 (6.20) |
  Day 168: number analyzed (Participants) | 29 | 0
  Day 168 | 27.5 (8.37) |
  Day 252: number analyzed (Participants) | 26 | 0
  Day 252 | 31.0 (11.2) |
  Day 308: number analyzed (Participants) | 26 | 0
  Day 308 | 29.9 (11.0) |
  Day 336: number analyzed (Participants) | 25 | 0
  Day 336 | 27.8 (10.9) |

5. Secondary Outcome: Maximum Observed Serum Concentration(Cmax) Derived on Day 1, 168 and 308
Description: Cmax is the observed maximum plasma concentration following administration (μg/mL).
Time Frame: Day 1, 168, 308 at pre-dose and 45 mins post-dose
Population: Pharmacokinetics (PK) analysis set - PK samples were only obtained and evaluated for subjects treated with BYM338
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | BYM338 10 mg/kg | Placebo
Number analyzed (Participants) | 36 | 0
μg/mL
  Day 1 | 283 (32.0) |
  Day 168: number analyzed (Participants) | 29 | 0
  Day 168 | 292 (45.3) |
  Day 308: number analyzed (Participants) | 27 | 0
  Day 308 | 271 (31.1) |

6. Secondary Outcome: Time to Reach the Maximum Concentration After Drug Administration (Tmax) Derived on Day 168 and 308
Description: Tmax is the time to reach peak or maximum concentration (h) after the drug administration.
Time Frame: Day 1, 168, 308 at pre-dose and 45 mins post-dose
Population: Pharmacokinetics (PK) analysis set - PK samples were only obtained and evaluated for subjects treated with BYM338
Measure: Median (Inter-Quartile Range); unit: hr
Arm/Group | BYM338 10 mg/kg | Placebo
Number analyzed (Participants) | 36 | 0
hr
  Day 1 | 0.750 [0.683 to 0.917] |
  Day 168: number analyzed (Participants) | 29 | 0
  Day 168 | 0.750 [0.750 to 1.05] |
  Day 308: number analyzed (Participants) | 27 | 0
  Day 308 | 0.750 [0.750 to 1.38] |

7. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Body Mass Index (BMI) was determined by height and weight measurements at week 24 and 48. A negative change from baseline indicates improvement. BMI was calculated as (Body weight (kg)/ [Height (m)]^2)
Time Frame: Baseline, Week 24, Week 48
Population: Pharmacodynamic analysis set
Measure: Least Squares Mean (80% Confidence Interval); unit: Kg/m^2
Arm/Group | BYM338 10 mg/kg | Placebo
Number analyzed (Participants) | 36 | 36
Kg/m^2
  week 24: number analyzed (Participants) | 29 | 31
  week 24 | -1.50 [-1.77 to -1.23] | -0.17 [-0.43 to 0.10]
  week 48: number analyzed (Participants) | 26 | 30
  week 48 | -2.19 [-2.60 to -1.78] | -0.28 [-0.67 to 0.11]
Statistical Analysis 1: Comparison: BYM338 10 mg/kg vs Placebo; week 24; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = -1.33, 80% CI 2-sided [-1.71 to -0.95]
Statistical Analysis 2: Comparison: BYM338 10 mg/kg vs Placebo; week 48; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = -1.91, 80% CI 2-sided [-2.48 to -1.34]

8. Secondary Outcome: Change From Baseline in Weight
Description: Body weight was measured to the nearest 0.1 kilogram (kg) in indoor clothing without shoes. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 24, Week 48
Population: Pharmacodynamic analysis set
Measure: Least Squares Mean (80% Confidence Interval); unit: Kg
Arm/Group | BYM338 10 mg/kg | Placebo
Number analyzed (Participants) | 36 | 36
Kg
  week 24: number analyzed (Participants) | 29 | 31
  week 24 | -3.99 [-4.79 to -3.19] | -0.57 [-1.34 to 0.21]
  week 48: number analyzed (Participants) | 26 | 30
  week 48 | -5.90 [-7.08 to -4.71] | -0.79 [-1.92 to 0.33]
Statistical Analysis 1: Comparison: BYM338 10 mg/kg vs Placebo; week 24; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = -3.43, 80% CI 2-sided [-4.54 to -2.31]
Statistical Analysis 2: Comparison: BYM338 10 mg/kg vs Placebo; week 48; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = -5.10, 80% CI 2-sided [-6.74 to -3.47]

9. Secondary Outcome: Change From Baseline in Lean Body Mass (LBM) Measured by DXA
Description: Lean body mass (LBM) is a part of body composition defined as the difference between total body weight and body fat weight. This means that it counts the mass of all organs except body fat, including bones, muscles, blood, skin, and everything else.
  Dual energy X-ray absorptiometry (DXA) was used to assess changes in body composition, including total fat and lean body mass (FM and LBM) and appendicular skeletal fat and muscle mass (aFM and aLBM). DXA instruments had a source that generated x-rays split into two energies which measured bone mineral mass and soft tissue from which fat and fat-free mass (or lean body mass) were estimated.
Time Frame: Baseline, Week 24, Week 48
Population: Pharmacodynamic analysis set
Measure: Least Squares Mean (80% Confidence Interval); unit: Kg
Arm/Group | BYM338 10 mg/kg | Placebo
Number analyzed (Participants) | 36 | 36
Kg
  week 24: number analyzed (Participants) | 29 | 31
  week 24 | 1.72 [1.25 to 2.19] | 0.23 [-0.23 to 0.68]
  week 48: number analyzed (Participants) | 26 | 29
  week 48 | 1.70 [1.14 to 2.26] | -0.44 [-0.97 to 0.09]
Statistical Analysis 1: Comparison: BYM338 10 mg/kg vs Placebo; week 24; Test type: Superiority; p = 0.003, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = 1.49, 80% CI 2-sided [0.82 to 2.06]
Statistical Analysis 2: Comparison: BYM338 10 mg/kg vs Placebo; week 48; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = 2.14, 80% CI 2-sided [1.36 to 2.93]

10. Secondary Outcome: Change From Baseline in Waist Circumference
Description: Waist circumference is the length in cm of the circumference to the nearest 0.1 cm at the level of the umbilicus with the subject in the upright position. A negative change indicates improvement.
Time Frame: Baseline, Week 24, Week 52
Population: Pharmacodynamic analysis set
Measure: Least Squares Mean (80% Confidence Interval); unit: cm
Arm/Group | BYM338 10 mg/kg | Placebo
Number analyzed (Participants) | 36 | 36
cm
  week 24: number analyzed (Participants) | 29 | 31
  week 24 | -5.04 [-5.87 to -4.20] | -0.95 [-1.75 to -0.14]
  week 52: number analyzed (Participants) | 26 | 30
  week 52 | -9.00 [-10.3 to -7.68] | 0.45 [-0.79 to 1.69]
Statistical Analysis 1: Comparison: BYM338 10 mg/kg vs Placebo; week 24; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = -4.09, 80% CI 2-sided [-5.26 to -2.92]
Statistical Analysis 2: Comparison: BYM338 10 mg/kg vs Placebo; week 52; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = -9.46, 80% CI 2-sided [-11.3 to -7.64]

11. Secondary Outcome: Change From Baseline in Waist to Hip Ratio
Description: Hip circumference was measured at the greatest protrusion of the buttocks. Combined with waist circumference, the waist-to-hip ratio was derived during data analysis.
Time Frame: Baseline, Week 24, Week 52
Population: Pharmacodynamic analysis set
Measure: Least Squares Mean (80% Confidence Interval); unit: ratio
Arm/Group | BYM338 10 mg/kg | Placebo
Number analyzed (Participants) | 36 | 36
ratio
  week 24: number analyzed (Participants) | 29 | 31
  week 24 | -0.02 [-0.03 to -0.01] | -0.01 [-0.01 to 0.00]
  week 52: number analyzed (Participants) | 26 | 30
  week 52 | -0.05 [-0.06 to -0.04] | 0.01 [0.00 to 0.02]
Statistical Analysis 1: Comparison: BYM338 10 mg/kg vs Placebo; week 24; Test type: Superiority; p = 0.062, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = -0.02, 80% CI 2-sided [-0.03 to -0.00]
Statistical Analysis 2: Comparison: BYM338 10 mg/kg vs Placebo; week 52; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = -0.06, 80% CI 2-sided [-0.08 to -0.04]

12. Secondary Outcome: Change From Baseline in Insulin Resistance (HOMA2-IR)
Description: Blood samples were collected to analyze insulin resistance. The homeostasis model assessment computational method was used to estimate insulin resistance (HOMA2-IR) from fasting plasma glucose and insulin. The HOMA2-IR is the reciprocal of insulin sensitivity (%S), as a percentage of a normal reference population (normal young adult). Higher numbers indicate higher insulin resistance. No established cutoffs are indicating impaired resistance. HOMA2-IR was calculated using an online calculator [https://www.dtu.ox.ac.uk/homacalculator/].
Time Frame: Baseline. Week 12, Week 36
Population: Pharmacodynamic analysis set
Measure: Least Squares Mean (80% Confidence Interval); unit: Insulin Resistance (IR) Score
Arm/Group | BYM338 10 mg/kg | Placebo
Number analyzed (Participants) | 36 | 36
Insulin Resistance (IR) Score
  week 12: number analyzed (Participants) | 29 | 31
  week 12 | 0.10 [-0.17 to 0.37] | 0.76 [0.50 to 1.02]
  week 36: number analyzed (Participants) | 25 | 27
  week 36 | -0.09 [-0.44 to 0.25] | 0.57 [0.24 to 0.90]
Statistical Analysis 1: Comparison: BYM338 10 mg/kg vs Placebo; week 12; Test type: Superiority; p = 0.028, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = -0.65, 80% CI 2-sided [-1.03 to -0.28]
Statistical Analysis 2: Comparison: BYM338 10 mg/kg vs Placebo; week 36; Test type: Superiority; p = 0.081, Mixed-Effect Model Repeated Measure; Mean Difference (Net) = -0.66, 80% CI 2-sided [-1.14 to -0.18]

13. Secondary Outcome: Immunogenicity Assessed by the Number of Participants Developing Anti-BYM338 Antibodies During the Trial
Description: Describes the number of participants tested positive for anti-BYM338 antibodies after the start of bimagrumab (BYM338) treatment. A validated bridging enzyme-linked immunosorbent assay (ELISA) was used for the confirmation of the presence of anti-BYM338 antibodies in human serum.
Time Frame: 392 days
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BYM338 10 mg/kg | Placebo
Number analyzed (Participants) | 37 | 38
Participants
  Confirmed with positive immunogenicity | 2 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study for 56 weeks which includes the treatment period of 48 weeks and the follow-up period of 8 weeks.
Arm/Group | BYM338 10 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 3/37 | 3/38
Other Adverse Events (participants affected / at risk) | 31/37 | 31/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338 10 mg/kg (N=37) | Placebo (N=38)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Lipase increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338 10 mg/kg (N=37) | Placebo (N=38)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Thyroid cyst (Endocrine disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0
Macular oedema (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 15 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Early satiety (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Influenza like illness (General disorders) | 0 | 1
Infusion site extravasation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 2
Sialoadenitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0
Amylase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 4 | 2
Pancreatic enzymes increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 5
Paraesthesia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 1
Phlebitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT03005288/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT03005288/SAP_001.pdf